CLINICAL TRIAL: NCT00000417
Title: A Randomized Controlled Trial of a Psychoeducational Intervention to Improve Outcomes in Systemic Lupus Erythematosus (SLE)
Brief Title: Psychoeducational Approach to Improve Health in Lupus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Matthew H. Liang, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P60 AR36308 NIAMS-014; P60AR036308 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Educational intervention; Health education; Social support network; Outcomes research; Self-help
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Health Education | interventions — Counseling

INTERVENTIONS:
Procedure: Counseling intervention
Device: Informational film

SUMMARY:
We will study the relationships among patient/partner communication, social support, and self-efficacy (a person's belief in the ability to manage his or her disease) as they affect the health of people with systemic lupus erythematosus (SLE, or lupus) over time. We are assigning 150 people with lupus and their partners to either (1) receive counseling to improve self-efficacy, partner support, and patient/partner problem solving or (2) see an informational film about lupus. We will follow study participants for 12 months to find out about their physical and mental health, disease activity, beliefs that they can take steps that help them feel better, coping, social support, and couples communication.

DETAILED DESCRIPTION:
Studies have shown that patient self-efficacy in disease management and social support predict physical and mental health and disease activity in lupus. We wished to study the relationships among patient/partner communication, social support, and self-efficacy as they influence patient health longitudinally. We are randomizing 150 lupus patients and their partners to either (1) participate in a counseling intervention to improve self-efficacy, partner support, and patient/partner problem-solving in lupus management or (2) see an informational film about lupus (control). The counseling intervention includes an initial in-person session followed by five monthly telephone calls to monitor and reinforce problem-solving. We will follow patients for 12 months for self-reported physical and mental health, disease activity, self-efficacy, coping, social support, and couples communication.

ELIGIBILITY:
Inclusion Criteria:

* Has partner willing to participate in study

Exclusion Criteria:

* Unable to read and write English questionnaires
* Unable to be reached by phone
* Rheumatologist considers patient unable to participate, generally due to patient cognitive problems or severe illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1997-04; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawren H. Daltroy, DrPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Karlson EW, Liang MH, Eaton H, Huang J, Fitzgerald L, Rogers MP, Daltroy LH. A randomized clinical trial of a psychoeducational intervention to improve outcomes in systemic lupus erythematosus. Arthritis Rheum. 2004 Jun;50(6):1832-41. doi: 10.1002/art.20279. PMID 15188360